CLINICAL TRIAL: NCT05922215
Title: Effects of Balance Training on Gait and Functional Strength in Children With Intellectual Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/0707
Record Dates: First submitted 2023-03-15; First posted 2023-06-28 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Intellectual Impairment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Other: Dynamic Balance training; Other: Static balance training
- Control Group (Active Comparator)
  Interventions: Other: Static balance training

INTERVENTIONS:
Other: Dynamic Balance training — The Experimental group will be given the Baseline treatment comprising of Stretching & Static balance training (i.e. heel and toe raises, alternate rising of the left and right foot above the floor and tandem standing.) alongside Dynamic Balance training which will include (weight shifting forward, backward, sideward, and diagonally with eyes opened and eyes closed, walking toe-to-heel barefoot, side walking, reverse walking and one-foot jumps), and Progressive activity training (such as stepping over/on obstacles, throwing and catching a ball, and kicking a ball.) for 40 minutes per day, twice each week for 8 weeks.
  Arms: Experimental Group
Other: Static balance training — The Control group will continue their regular school schedule, which will include participation in physical education activities at the same frequency. Along with that Baseline treatment including Static balance training (i.e. alternate rising of the left and right foot above the floor and tandem standing.) only, at the same intervals and for the same length of time as the intervention group, with the exception of additional Dynamic balance training and progressive activity training.

SUMMARY:
Intellectual impairment is a developmental condition that first appears in childhood and causes substantial intellectual or cognitive limitations as well as inadequate adaptation to the demands of daily life. It may be viewed as a syndrome grouping (meta-syndrome), rather than as an illness or a disability; encompassing a wide range of clinical problems, including hereditary, viral, metabolic, and neurological issues. Prior to learning new abilities, there is a loss in cognitive functioning that is indicative of ID. Falling is a severe issue that affects people with intellectual disabilities frequently. Although studies based on retrospective data collected over time have not determined the exact prevalence of falling in the ID community, they have estimated that 30-60% of people fall within a 12-month period. Similar fall risk factors exist in the general population and in people with ID, such as advancing age, vision problems, and mobility issues. However, some characteristics, such as having frequent seizures and a high level of ambulation, seem more distinctive to ID. The purpose of this study is to analyze the effects of balance training on gait and functional strength in children with mild intellectual disabilities. This will be a Randomized Controlled Trial. Approval will be gained from the Ethical committee of the Riphah international university Lahore, Pakistan prior to the commencement of study. Written informed consent will be taken from all the patients and all information and data will be confidential. Subjects will be informed that there is no risk of study and they will be free to withdraw any time during process of study. 22 intellectually disabled children between the ages of 7 and 14 will be randomly allocated to the Experimental group (n=10) or a Control group (n=10). The Experimental group will be given the Baseline treatment comprising of Static balance training (i.e. heel and toe raises, alternate rising of the left and right foot above the floor and tandem standing.) alongside Dynamic Balance training (weight shifting forward, backward, sideward, and diagonally with eyes opened and eyes closed, walking toe-to-heel barefoot, side walking, reverse walking and one-foot jumps), and Progressive activity training (including stepping over/on obstacles, throwing and catching a ball, and kicking a ball.) for 40 minutes per day, twice each week for 8 weeks. Whereas, the Control group will continue their regular school schedule, which will include participation in physical education activities at the same frequency. Along with that, only Baseline treatment including Static balance training (i.e. alternate rising of the left and right foot above the floor and tandem standing.) will be given at the same intervals and for the same length of time as the intervention group, with the exception of additional Dynamic balance training and progressive activity training. The time up-and-go test, the 10-meter walk test and GMFM-88 were used to evaluate gait, and the Sit-to-stand test and the Stair Climbing test. were used to measure each participant's functional strength. Pre and Post treatment values will be evaluated and the Data will be analyzed using SPSS 22.0.

ELIGIBILITY:
Inclusion Criteria:

* Boys and Girls with Mild Intellectual Disabilities (IQ range 50-69)
* Age group: 7-14 years
* Students from a Special Education School

Exclusion Criteria:

* CP and Down's syndrome
* Those who were unable to complete follow-up tests.
* Subjects who took part in less than 80% of the intervention program.
* Participants with any psychological or behavioral issues.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Time Up and Go test | Baseline and 8th week
  The Time Up and Go test (TUG) is a quick test that measures balance in both the static and dynamic planes. It uses the time that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees. During the test, the person is expected to wear their regular footwear and use any mobility aids that they would normally require.
Change in Sit to stand test | Baseline and 8th week
  The Sit to stand also known as the 30 Second Chair Stand Test (30CST) is administered to test leg strength and endurance. Equipment: A chair with a straight back without arm rests (seat 17" high), and a stopwatch.
  Method: The participant is urged to complete as many full stands as they can in the allotted 30 seconds. Between each stand, the person is told to sit down completely. The tester silently counts the completion of each correct stand while keeping an eye on the participant's performance to verify perfect form.
Change in Stair climb test | baseline and 8th week
  The stair climb test, also known as the stair climb power test, is a field-based evaluation of lower body strength, power, and physical function that is clinically relevant, safe, and affordable. Equipment: Stairs (8 - 14 steps) with handrails, stopwatch. Scoring: Total time to ascend and descend steps is recorded to the nearest 100th of a second.
  The patient should use the assistive device (if any) normally used to perform the activity at the time of testing.

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Rising Sun Institute for special children, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vuijk PJ, Hartman E, Scherder E, Visscher C. Motor performance of children with mild intellectual disability and borderline intellectual functioning. J Intellect Disabil Res. 2010 Nov;54(11):955-65. doi: 10.1111/j.1365-2788.2010.01318.x. Epub 2010 Sep 20. PMID 20854287
- [Background] Wang J, Gao Y, Kwok HHM, Huang WYJ, Li S, Li L. Children with Intellectual Disability Are Vulnerable to Overweight and Obesity: A Cross-Sectional Study among Chinese Children. Child Obes. 2018 Jul;14(5):316-326. doi: 10.1089/chi.2018.0015. Epub 2018 Jul 5. PMID 29975552
- [Background] Stanish HI, Curtin C, Must A, Phillips S, Maslin M, Bandini LG. Physical Activity Enjoyment, Perceived Barriers, and Beliefs Among Adolescents With and Without Intellectual Disabilities. J Phys Act Health. 2016 Jan;13(1):102-10. doi: 10.1123/jpah.2014-0548. Epub 2015 Apr 1. PMID 25830443
- [Background] Maiano C, Hue O, Morin AJS, Lepage G, Tracey D, Moullec G. Exercise interventions to improve balance for young people with intellectual disabilities: a systematic review and meta-analysis. Dev Med Child Neurol. 2019 Apr;61(4):406-418. doi: 10.1111/dmcn.14023. Epub 2018 Sep 19. PMID 30230530